CLINICAL TRIAL: NCT07002502
Title: Immune Modulation and Efficacy Assessment of PRaG-1 in Patients With Advanced Solid Malignancies: A Prospective, Multicenter, Open-Label Clinical Trial
Brief Title: Immune Modulation With PRaG-1 Treatment
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Second Affiliated Hospital of Soochow University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LK2025016
Record Dates: First submitted 2025-05-25; First posted 2025-06-03 (Actual); Last update posted 2025-06-10 (Actual); Status verified 2025-05

CONDITIONS: Cancer; Solid Cancer
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- PRaG-1 treatment (Experimental)
  Interventions: Drug: PRaG-1(cordycepin tablet)

INTERVENTIONS:
Drug: PRaG-1(cordycepin tablet) — The "PRaG-1" cordycepin tablet involved in this clinical study is produced by Shengmingyuan Company, a subsidiary of the National Biochemical Engineering Research Center at Nanjing Tech University. It is an oral tablet, with each tablet containing 200 mg of cordycepin. The product has obtained a national food production license, and the production license number is SC11332019200201.

SUMMARY:
The study is a single-center, prospective, single-arm, Phase II clinical trial. Eligible patients with advanced solid malignant tumors will sign the informed consent form and undergo screening for enrollment. After enrollment, patients will receive oral administration of "PRaG-1" twice daily (morning and evening) for a total of 10 days. Peripheral blood lymphocyte tests will be performed before treatment, on day 5 post-treatment, and at the conclusion of treatment.

DETAILED DESCRIPTION:
The "PRaG-1" cordycepin tablet involved in this clinical study is produced by Shengmingyuan Company, a subsidiary of the National Biochemical Engineering Research Center at Nanjing Tech University. It is an oral tablet, with each tablet containing 200 mg of cordycepin. The product has obtained a national food production license, and the production license number is SC11332019200201.

Patients will receive "PRaG-1" treatment twice daily (morning and evening) for a total of 10 days. Peripheral blood lymphocyte tests will be performed at pre-treatment, after 5 days of treatment, and at the end of treatment. A 5 ml blood sample and 2 g of tissue will be collected via biopsy before and after treatment for storage, to be used in subsequent analysis of immune function-related indicators. The clinical trial will be terminated if any of the following occur: disease progression, intolerable toxicity, withdrawal of the informed consent form (ICF), death, or other conditions specified in the protocol that require discontinuation of treatment.

ELIGIBILITY:
Inclusion Criteria:

Patients with a history of other malignant diseases within the past 5 years, except for curatively treated skin cancer and cervical carcinoma in situ; Patients with a history of uncontrolled epilepsy, central nervous system diseases, or psychiatric disorders, which, in the judgment of the investigator, may impair the ability to sign the informed consent form or affect the patient's compliance with drug treatment; Clinically significant (i.e., active) cardiovascular disease, such as symptomatic coronary artery disease, New York Heart Association (NYHA) Class II or worse congestive heart failure, or severe arrhythmias requiring medication, or a history of myocardial infarction within the past 12 months; Patients currently receiving immunosuppressive therapy; Known active major infections, or significant hematological, renal, metabolic, gastrointestinal, endocrine dysfunction, or other serious uncontrolled comorbid conditions, as determined by the investigator; Patients with hypersensitivity to any component of the investigational drugs; History of immunodeficiency, including positive HIV test results or other acquired or congenital immunodeficiency diseases, history of organ transplantation, or other immunologically related conditions requiring long-term oral steroid therapy; Other conditions deemed unsuitable for enrollment by the investigator.

Exclusion Criteria:

Patients with a history of any other malignant diseases within the past 5 years are excluded, except for curatively treated skin cancer and cervical carcinoma in situ.

Patients with a history of uncontrolled epilepsy, central nervous system diseases, or psychiatric disorders are excluded if, in the judgment of the investigator, these conditions may impair the ability to sign the informed consent form or affect the patient's compliance with drug treatment.

Clinically significant (active) cardiovascular disease is excluded, including symptomatic coronary artery disease, New York Heart Association (NYHA) Class II or worse congestive heart failure, severe arrhythmias requiring medication, or a history of myocardial infarction within the past 12 months.

Patients currently receiving immunosuppressive therapy are excluded. Known active major infections are excluded, as are significant hematological, renal, metabolic, gastrointestinal, endocrine dysfunction, or other serious uncontrolled comorbid conditions, as determined by the investigator.

Patients with hypersensitivity to any component of the investigational drugs are excluded.

History of immunodeficiency is excluded, including positive HIV test results, other acquired or congenital immunodeficiency diseases, history of organ transplantation, or other immunologically related conditions requiring long-term oral steroid therapy.

Other conditions deemed unsuitable for enrollment by the investigator are excluded.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 19 (Estimated)
Dates: Start 2025-06-15 (Estimated); Primary Completion 2026-05-26 (Estimated); Study Completion 2026-06-26 (Estimated)

PRIMARY OUTCOMES:
Peripheral blood lymphocyte subsets | 10 days
  the change of peripheral blood lymphocyte subsets

SECONDARY OUTCOMES:
Adverse event | 3 months
  rate of adverse events